CLINICAL TRIAL: NCT05447156
Title: QuitGuide for American Indians: Aims 2 & 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-2022-30604; MCC CPRC (Other: 2022LS018)
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Aim 3: Participants will be randomized to either the tailored QuitGuide app or the standard version of the QuitGuide app for 5 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 3:Tailored App (Experimental): Randomized subset of participants will use the tailored QuitGuide app, a smoking cessation app, downloaded to their personal phone.
  Interventions: Behavioral: Tailored QuitGuide app
- Aim 3: Standard App (Placebo Comparator): Randomized subset of participants will use the standard QuitGuide app, a smoking cessation app available to the public, downloaded to their personal phone.
  Interventions: Behavioral: Standard QuitGuide app

INTERVENTIONS:
Behavioral: Tailored QuitGuide app — This is an app not available to the public. It was developed/tailored based on an app available to the public and can be downloaded.
  Arms: Aim 3:Tailored App
Behavioral: Standard QuitGuide app — This is an app available to the public.
  Arms: Aim 3: Standard App

SUMMARY:
Aim 3: To test feasibility, acceptability, and preliminary efficacy of the tailored QuitGuide for smoking cessation among AIs.

ELIGIBILITY:
Inclusion Criteria:

* American Indian person based on self-report
* Age ≥ 18 years
* Interested in quitting smoking
* Smoke ≥ 3 commercial tobacco cigarette per day (CPD) in the past 30 days

  o Use of other commercial tobacco products (e.g., e-cigarettes) is permitted if they report cigarettes being their primary product
* Smartphone ownership with the ability to download applications and sufficient data to complete research procedures

Exclusion Criteria:

* New or change in pharmacotherapy for smoking cessation (includes: nicotine gum, patch, lozenge, inhaler OR medications Chantix/Wellbtrutin/Zyban/Bupropion) in past month
* Does not speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Caroll, PhD, Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota
Locations (1):
- Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Started | 58 | 57
Completed | 55 | 53
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  >18 years | 58 | 57 | 115
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex not reported for one participant.
  Participants
    number analyzed (Participants) | 57 | 57 | 114
    Female | 46 | 42 | 88
    Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 56 | 55 | 111
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 52 | 51 | 103
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 115

OUTCOME MEASURES:

1. Primary Outcome: Frequency of App Use
Description: The number of times the app is initiated per day will be measured using data from Smokefree.gov. If a participant does not use the app on a particular day, Smokefree.gov records this as non-use or 0 for that day. The total number of times will be summarized for analysis by totaling the number of times the app is initiated from randomization to 5 weeks post-randomization.
Time Frame: 5 weeks post enrollment and 1 week post randomization
Measure: Mean (Standard Deviation); unit: App initiations per day
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Number analyzed (Participants) | 58 | 57
App initiations per day
  5 weeks post enrollment | 15.3 (15.5) | 14.9 (17.8)
  1 week post randomization | 4.3 (5.1) | 3.7 (3.6)

2. Secondary Outcome: Study Attrition Measured as Percentage of Randomized Participants That Complete the Final Phone Interview at 5 Weeks
Description: Percentage of randomized participants that complete the final phone interview at 5 weeks
Time Frame: 5 weeks post enrollment aim 3
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Number analyzed (Participants) | 58 | 57
Participants | 55 | 53

3. Secondary Outcome: Frequency of Returning Saliva Sample by 2 Weeks Post the Week 5 Interview
Description: Count of randomized participants that return saliva sample 2 weeks after the 5 weeks post enrollment (end of intervention)
Time Frame: 5 weeks post enrollment aim 3
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Number analyzed (Participants) | 58 | 57
Participants | 35 | 31

4. Secondary Outcome: Usability of App Design Measured Using System Usability Scale (SUS)
Description: Scores for each question (1-5) are added together for an overall score of 100. 100 means the website is rated at optimal usability. Scores lower than 100 indicate the website needs improvements. Mean and standard deviations or medians and ranges of percentile rankings will be calculated. Minimum score of zero.
Time Frame: 5 weeks post enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Number analyzed (Participants) | 55 | 53
score on a scale | 72.4 (15.6) | 71.9 (13.3)

5. Secondary Outcome: Acceptability of Overall App
Description: Mean and standard deviations or medians and ranges of Likert-scale responses to questions such as 'How likely would you be to recommend the app to a friend?'. Rated out of 7 points. 7 is the highest score, indicating participants are very likely to recommend the app to a friend. Scores lower than 7 indicate participants are less likely to recommend the app. Minimum score of zero.
Time Frame: 5 weeks post enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Number analyzed (Participants) | 55 | 53
units on a scale | 5.6 (1.6) | 4.9 (1.6)

6. Secondary Outcome: Fit of App With Culture
Description: Mean and standard deviations or medians and ranges of Likert-scale responses to questions such as 'The app fits my American Indian culture such as its history, traditions, and customs'. Rated out of 7 points. 7 is the highest score, indicating participants feel app fits the American Indian culture. Scores lower than 7 indicate participants don't feel as strongly that app fits American Indian culture. Minimum score of zero.
Time Frame: 5 weeks post enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
Number analyzed (Participants) | 55 | 53
units on a scale | 3.9 (0.9) | 3.1 (1.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aim 3:Tailored App | Aim 3: Standard App
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 0/58 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05447156/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT05447156/ICF_000.pdf